CLINICAL TRIAL: NCT05706922
Title: Changes in the Gut- and Vaginal Microbiome Composition in Association With PCOS Clinical Phenotypes.
Brief Title: Gut- and Vaginal Microbiome Composition in Association With PCOS
Acronym: GuVaPCOS
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Sam Schoenmakers, Principal Investigator, Erasmus Medical Center
Other Study IDs: NL80648.078.22
Record Dates: First submitted 2023-01-11; First posted 2023-01-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: gut microbiome; vaginal microbiome; polycystic ovary syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Polycystic ovary syndrome (PCOS): * Hormonal screening
  * Vaginal swab
  * Fecal sample
  * Blood samples
  * Food Frequency Questionnaire
  Interventions: Other: Venous blood sample, vaginal swab
- Control group: * Hormonal screening
  * Vaginal swab
  * Fecal sample
  * Blood samples
  * Food Frequency Questionnaire
  Interventions: Other: Venous blood sample, vaginal swab

INTERVENTIONS:
Other: Venous blood sample, vaginal swab — Venous blood samples and vaginal swab will be obtained on the same day.

SUMMARY:
Polycystic ovary syndrome (PCOS) is an endocrine disorder that affects up to 10% of the reproductive-aged women worldwide. The etiology is still unknown and treatment therefore remains symptomatic. Studies indicate a possible role of the gut microbiome in the pathology of PCOS. PCOS women have a disturbed gut microbiome, with certain species associated with the PCOS characteristics:hyperandrogenism, ovarian dysfunction, obesity, glucose intolerance and insulin resistance. Although differences have been found in gut microbiome composition between PCOS and healthy women, the literature is inconclusive regarding the difference in gut microbiome biodiversity. Studies examining the vaginal microbiome in PCOS women show consistent results with specific species in the vaginal microbiome. However, there are only few studies on the vaginal microbiome in PCOS women and no studies have yet investigated the correlation between sex-specific hormones and PCOS characteristics. More research is needed to understand the function of the microbiome in the pathophysiology of PCOS, so that this can offer perspectives in future therapies.

ELIGIBILITY:
Inclusion criteria

* Caucasian
* Willing to provide vaginal swab and stool sample
* Willing to provide informed consent
* Sufficient command of the Dutch language
* Diagnosed with PCOS at Erasmus MC using the Rotterdam criteria by the presence of at least two of the following criteria
* Clinical or biochemical hyperandrogenism (modified Ferriman-Gallway score >5; testosterone level >2nmol/L, Free Androgen Index > 2.9)
* Oligomenorrorrhea or amenorrhea
* Polycystic ovaries.

Exclusion criteria

* BMI <18
* Smoking
* Diabetes Mellitus or use of insulin sensitizer
* Chronic and acute infection diseases
* Endometriosis (American Fertility Score (AFS) III/IV)
* Elevated prolactin levels, thyroid disease, Cushing disease or gastro-intestinal disease
* The use of hormonal contraceptives, and other steroid hormones in the last 3 months
* Use of antibiotics, probiotics or laxatives in the last 3 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients at the outpatient clinic of Reproductive Medicine.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Bacterial composition of the gut in women with PCOS and control group | 1 week
  Bacterial composition in the gut is analysed using 16S rRNA gene sequencing

SECONDARY OUTCOMES:
Bacterial composition of the vagina in women with PCOS and control group | 1 week
  Bacterial composition in the vagina is analysed using 16S rRNA gene sequencing
Difference in bacterial composition of the vagina and gut in women with PCOS | 1 week
  Relative abundance of bacterial communities
Difference in bacterial composition of the vagina and gut between overweight/obese and lean patients (with/without PCOS) | 1 week
  Relative abundance of bacterial communities
To analyse potential metabolic profiles characterizing different phenotypes of PCOS | 1 week
  Expression of metabolic indicators (metabolomics)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Schoenmakers, Dr. drs., Principal Investigator — Division of Obstetrics and Fetal Medicine, Department of Obstetrics and Gynecology; Joop S.E. Laven, Prof. dr., Study Director — Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology
Locations (1):
- Erasmus University Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT05706922/Prot_000.pdf